CLINICAL TRIAL: NCT01272336
Title: Intermittent Hypoxia Promotes Restoration of Hand Function Following SCI
Brief Title: Study Effects of Intermittent Hypoxia on Restoring Hand Function Following SCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of Saskatchewan (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Randy D. Trumbower, Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00035986; 163907 (Other: Other)
Record Dates: First submitted 2011-01-04; First posted 2011-01-07 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury, low oxygen, strength, motor control
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIH/Sham (Active Comparator): Subjects with chronic, motor-incomplete SCI receive AIH and then SHAM
  Interventions: Drug: Acute Intermittent Hypoxia (AIH); Other: SHAM-Intermittent Room Air
- Sham/AIH (Active Comparator): Subjects with chronic, motor-incomplete SCI receive SHAM and then AIH
  Interventions: Drug: Acute Intermittent Hypoxia (AIH); Other: SHAM-Intermittent Room Air

INTERVENTIONS:
Drug: Acute Intermittent Hypoxia (AIH) — Participants will breath intermittent low oxygen via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of FIO2=0.09±0.02 (hypoxia) air for 15 minutes.Participants will receive treatment for up to seven visits.
  Other Names: Hypoxia air mixture
Other: SHAM-Intermittent Room Air — This is a sham intervention to the AIH intervention. Participants will breath intermittent room air via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of FIO2=0.21±0.02 (normoxia). Participants will receive treatment for up to seven visits.
  Other Names: Room air mixture

SUMMARY:
The goal of the study is to examine the effects of repeated breathing episodes of mild intermittent hypoxia (reduced oxygen) training on hand strength and grasping ability following cervical spinal injury, and to determine whether these changes result in improved hand function. If so, such changes may indicate hypoxia-induced spinal plasticity (ability of the nervous system to strengthen neural pathways based on new experiences), which could result in improvements in hand use for persons with spinal cord injury (SCI).

DETAILED DESCRIPTION:
The goal of the study is to examine the effects of repeated breathing episodes of mild intermittent hypoxia (reduced oxygen) training on hand strength and grasping ability following cervical spinal injury, and to determine whether these changes result in improved hand function. If so, such changes may indicate hypoxia-induced spinal plasticity (ability of the nervous system to strengthen neural pathways based on new experiences), which could result in improvements in hand use for persons with spinal cord injury (SCI).

This idea stems from animal studies on respiration, in which investigators have shown that intermittent hypoxia induces spinal plasticity, strengthening neural connections within the spinal cord by a mechanism known as respiratory long-term facilitation. Exposure to mild hypoxia triggers oxygen sensors in the nervous system resulting in a cascade of events, including increased production of key proteins and, increased sensitivity of spinal cord circuitry necessary for improved respiration.

Because previous work using animal models has shown that similar events occur along non-respiratory pathways, the investigators propose to investigate whether a comparable dosing scheme of daily, mild intermittent hypoxia can positively affect upper limb function in persons with cervical SCI.

First, the investigators hypothesize that daily exposure of intermittent hypoxia training (7 consecutive days) will result in a sustained improvement in rat forelimb function that is dose-dependent. To test this hypothesis, the investigators will quantify the effects of variations in the number of intermittent hypoxia episodes on forelimb function in cervical spinal injured rats.

Second, the investigators hypothesize that daily exposure of intermittent hypoxia training will improve hand function in persons with cervical spinal injury. To test this hypothesis, the investigators will quantify the effect of mild intermittent hypoxia exposure, using a protocol derived from the animal model, on volitional grip strength and grasp function in persons with cervical SCI.

The effects of mild intermittent hypoxia, known to increase spinal motor activity, will be assessed as a possible therapeutic intervention to promote functionally useful hand recovery. Results from this study will be valuable for identifying novel strategies to control spinal neuron excitability and for improving motor function in persons with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and 65 years
* medical clearance to participate
* lesion below the 5th cervical spinous process (C5) and above the first thoracic spinous process (T1) with non-progressive etiology
* classified as motor-incomplete injury greater than 12 months
* independent breathing

Exclusion Criteria:

* Concurrent severe medical illness (i.e., infection, cardiovascular disease, ossification, recurrent autonomic dysreflexia, unhealed decubiti, and history of cardiac or pulmonary complications)
* Pregnant women because of the unknown affects of acute intermittent hypoxia on pregnant women and fetus
* Concomitant acquired brain injury
* History of seizures, brain injury, and/or epilepsy
* Diagnosed with obstructive sleep apnea
* Undergoing concurrent physical therapy
* Any contraindications to EMG testing procedures (skin sensitivity)
* Any contraindications to passive movement of the limbs
* Score of < 24 on Mini-Mental Exam

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Hand grasp | 1 week

SECONDARY OUTCOMES:
Grip strength | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Randy D Trumbower, PT, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Center for Rehabilitation Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Trumbower RD, Hayes HB, Mitchell GS, Wolf SL, Stahl VA. Effects of acute intermittent hypoxia on hand use after spinal cord trauma: A preliminary study. Neurology. 2017 Oct 31;89(18):1904-1907. doi: 10.1212/WNL.0000000000004596. Epub 2017 Sep 29. PMID 28972191